CLINICAL TRIAL: NCT07315373
Title: The FIND Study: A Dose-finding Study to Identify the Optimal Dose of Zanubrutinib in Adults With Immune Thrombocytopenia
Brief Title: Optimal Dose of Zanubrutinib to Treat Adult Immune Thrombocytopenia
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao Hui Zhang, Vice president of Peking University Institute of Hematology, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ITP-Find Study
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Immune Thrombocytopenia
Keywords: ITP; zanubrutinib
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — zanubrutinib; Dexamethasone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Zanubrutinib 80mg/d + Dexamethasone (Experimental): Participants in this arm will receive a combination therapy consisting of:
  Zanubrutinib: 80 mg taken orally once daily for 26 weeks. Dexamethasone: 40 mg taken orally once daily for 4 consecutive days at the beginning of treatment. A second identical 4-day course may be repeated after 2 weeks if an adequate initial platelet response is not achieved.
  Interventions: Drug: Zanubrutinib 80mg/d; Drug: High dose dexamethasone
- Zanubrutinib 160mg/d + Dexamethasone (Experimental): Participants in this arm will receive a combination therapy consisting of:
  Zanubrutinib: 160 mg taken orally once daily for 26 weeks. Dexamethasone: 40 mg taken orally once daily for 4 consecutive days at the beginning of treatment. A second identical 4-day course may be repeated after 2 weeks if an adequate initial platelet response is not achieved.
  Interventions: Drug: High dose dexamethasone; Drug: Zanubrutinib 160mg/d
- Zanubrutinib 240mg/d + Dexamethasone (Experimental): Participants in this arm will receive a combination therapy consisting of:
  Zanubrutinib: 240 mg taken orally once daily for 26 weeks. Dexamethasone: 40 mg taken orally once daily for 4 consecutive days at the beginning of treatment. A second identical 4-day course may be repeated after 2 weeks if an adequate initial platelet response is not achieved.
  Interventions: Drug: High dose dexamethasone; Drug: Zanubrutinib 240mg/d

INTERVENTIONS:
Drug: Zanubrutinib 80mg/d — Zanubrutinib: 80 mg taken orally once daily for 26 weeks
  Arms: Zanubrutinib 80mg/d + Dexamethasone
Drug: High dose dexamethasone — Dexamethasone: 40 mg taken orally once daily for 4 consecutive days at the beginning of treatment. A second identical 4-day course may be repeated after 2 weeks if an adequate initial platelet response is not achieved.
Drug: Zanubrutinib 160mg/d — Zanubrutinib: 160 mg taken orally once daily for 26 weeks
  Arms: Zanubrutinib 160mg/d + Dexamethasone
Drug: Zanubrutinib 240mg/d — Zanubrutinib: 240 mg taken orally once daily for 26 weeks
  Arms: Zanubrutinib 240mg/d + Dexamethasone

SUMMARY:
The goal of this clinical trial is to find the best dose of zanubrutinib when used together with high-dose dexamethasone for adults who are newly diagnosed with primary immune thrombocytopenia (ITP), and to learn how safe and effective this combination treatment is.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed newly-diagnosed, treatment-naive ITP;
2. Platelet counts <30×10^9/L ;
3. Platelet counts < 50×10^9/L and significant bleeding symptoms (WHO bleeding scale 2 or above);
4. Willing and able to sign written informed consent.

Exclusion Criteria:

1. Received chemotherapy or anticoagulants or other drugs affecting the platelet counts within 6 months before the screening visit;
2. Received first-line and second-line ITP-specific treatments (eg, steriods, cyclophosphamide, 6-mercaptopurine, vincristine, vinblastine, etc) ;
3. Current HIV infection or hepatitis B virus or hepatitis C virus infections;
4. Active infection;
5. Maligancy;
6. Severe medical condition (lung, hepatic or renal disorder) other than ITP. Unstable or uncontrolled disease or condition related to or impacting cardiac function (e.g., unstable angina, congestive heart failure, uncontrolled hypertension or cardiac arrhythmia);
7. Female patients who are nursing or pregnant, who may be pregnant, or who contemplate pregnancy during the study period; a history of clinically significant adverse reactions to previous corticosteroid therapy
8. Have a known diagnosis of other autoimmune diseases, established in the medical history and laboratory findings with positive results for the determination of antinuclear antibodies, anti-cardiolipin antibodies, lupus anticoagulant or direct Coombs test;
9. Patients who are deemed unsuitable for the study by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2028-12-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Sustained response | 26 weeks
  The maintenance of platelet count ≥ 30 x 10^9/L, at least 2-fold increase of the baseline count, the absence of bleeding, and no need for rescue medication at the 26-week follow-up.

SECONDARY OUTCOMES:
Initial Response (R) | day 14
  Response (R) as platelet count more than 30,000 per cubic millimeter and at least 2-fold increase of the baseline count and absence of bleeding.
Initial complete response (CR) | day 14
  Complete response (CR) was defined as platelet count more than 100,000 per cubic millimeter and absence of bleeding.
Time to response | 6 month
  The time from starting treatment to time of achievement of CR or R
Duration of response (DOR) | 26 weeks
  Duration of response at 26-week follow up
Bleeding events | 26 weeks
  Number of patients with bleeding
Adverse events | 26 weeks
  Number of patients with adverse events
Loss of response | 26 weeks
  Platelet counts below 100 x 109/L or bleeding (from CR) or platelet counts below 30 x 109/L, less than 2-fold increase of baseline platelet count or bleeding (from R)
Health related quality of life | baseline and 26 weeks
  Health-related quality of life using the Immune Thrombocytopenic Purpura-Patient Assessment Questionnaire (ITP-PAQ)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohui Zhang, Principal Investigator — Peking University People's Hospital, Peking University Institute of Hematology, National Clinical Research Center for Hematologic Disease, Beijing Key Laboratory of Hematopoietic Stem Cell Transplantation, Collaborative Innovation Center of Hematology

IPD SHARING:
Plan to Share IPD: Undecided